CLINICAL TRIAL: NCT02735447
Title: Pharmacoepidemiologic General Research Extension: PGRx-sIBM Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: La-ser Europe Limited (Other)
Responsible Party: Sponsor
Other Study IDs: LASER-PGRx
Record Dates: First submitted 2016-04-06; First posted 2016-04-12 (Estimated); Last update posted 2016-04-18 (Estimated); Status verified 2016-04

CONDITIONS: Sporadic Inclusion Body Myositis
MeSH Terms: conditions — Myositis, Inclusion Body

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Sporadic inclusion body myositis (sIBM) is a rare idiopathic inflammatory myopathy characterized by chronic proximal leg and distal arm asymmetric muscle weakness. Its prevalence is estimated between 10 and 100 cases per million, over the age of 50. Little is known about the natural course of the disease, the delay between onset and diagnosis, the patterns of disease management and treatment in routine practice, as well as the burden for patients.

The objectives of the PGRx-sIBM study will be to describe:

* The epidemiology of the disease (estimation of the prevalence, age at onset, delay between onset and diagnosis, diagnosis process, etc.)
* The patterns of disease management and treatment in routine practice
* The burden of the disease for patients and their informal caregiver, as well as the quality of life of patients
* The burden of the disease for informal caregivers

This will be an observational (non-interventional), cross-sectional (transversal) study.

Study setting The PGRx-sIBM will take place in France, Italy, Switzerland and Spain. Recruitment centers will be public and private practices and hospitals from urban or rural areas. In each recruitment center, at least one physician will act as a study investigator, in charge of identifying and recruiting patients.

Inclusion of patients

Patients will be included by their specialized physician (neurologist, Internal Medicine) during a regular outpatient visit, provided that they meet the following inclusion criteria:

* The patient has been diagnosed with sIBM, as per the physician judgement and regardless of the date of diagnosis
* Male or female
* Age ≥ 45 years old
* The patient does regularly live in the country of inclusion
* The patient or his/her proxy can read and respond to a telephone interview
* The patient agrees to participate

Exclusion criteria will be:

* The patient refuses to participate or the written Consent Form is not signed
* The patient or his/her proxy cannot be reached by telephone. All eligible patients will be invited to participate in the study, during a 3 to 6-month period of time.

The target sample size will be of 190 patients (≈15-20 in Switzerland, ≈50 in Spain, ≈50 in Italy and ≈70-75 in France).

ELIGIBILITY:
Inclusion Criteria:

* The patient has been diagnosed with sIBM, as per the physician judgement and regardless of the date of diagnosis
* Male or female
* Age ≥ 45 years old
* The patient does regularly live in the country of inclusion
* The patient or his/her proxy can read and respond to a telephone interview
* The patient agrees to participate

Exclusion Criteria:

* The patient refuses to participate or the written Consent Form is not signed
* The patient or his/her proxy cannot be reached by telephone.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with sporadic inclusion body myositis.
Sampling Method: Non-Probability Sample
Enrollment: 190 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-02 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Disability | Within the last 12 months
  Measured by the Clinical Global Impression scale and the use of assisitive devices
Quality of Life | Within the last 7 days
  EQ-D5

CONTACTS AND LOCATIONS:
Overall Officials: Lamiae Grimaldi-Bensouda, PharmD, PhD, Study Director — LASER